CLINICAL TRIAL: NCT07394413
Title: Surgical Handling of Fertility-preserving Treatments for Cervical Adenocarcinomas
Acronym: SHAFT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7939
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cervical Adenosarcoma
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite a growing body of literature on the subject, there is still uncertainty regarding direct comparisons between different conservative surgical techniques for cervical adenocarcinomas. In particular, it remains unclear whether fertility-sparing surgery for cervical adenocarcinomas - characterized by skip lesions - can ensure optimal disease control while achieving adequate obstetric outcomes.

For this reason, a systematic review and meta-analysis of the literature, along with an analysis of our center's data, is warranted. This approach will allow a critical, comparative evaluation of the efficacy of the different techniques (conization, simple trachelectomy, and radical trachelectomy) and the identification of prognostic factors to guide therapeutic choice.

ELIGIBILITY:
Inclusion Criteria:

* Adult women of reproductive age with a diagnosis of cervical adenocarcinoma
* Undergoing fertility-sparing surgery
* Minimum 12-month follow-up
* Signed informed consent

Exclusion Criteria:

* Histotypes other than cervical adenocarcinoma
* Undergoing radical surgery
* Follow-up less than 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women of reproductive age with cervical adenocarcinoma undergoing fertility-sparing surgery (conization, simple trachelectomy, radical trachelectomy) between 01/06/2019 and 30/06/2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 5 years
  The recurrence rate is defined as the proportion of patients who develop disease recurrence confirmed by imaging or histopathologic evaluation after FSS.
Disease free survival | 5 years
  Disease-free survival is defined as the time from surgery until the first documented recurrence.
Overall survival | 5 years
  Overall survival is measured as the time from surgery to death from any cause,

SECONDARY OUTCOMES:
pregnancy rate | 5 years
  Pregnancy rate is defined as the proportion of patients who achieve a clinically confirmed pregnancy among those attempting conception
live birth rate | 5 years
  Live birth rate is defined as the percentage of pregnancies that result in a live birth.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolò Bizzarri, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided